**COVER LETTER** 

We are writing to apply for NTC number for our project titled:

"Synergistic effect of Vitamin E and Vitamin D in reducing risk of side effects associated

typical anti-psychotics and improvement of psychiatric illness"

This particular research was designed as severe mental stress and psychotic illness are becoming

alarming and treatment therapy induces serious side effects like weight gain, change in lipid profile

and high blood pressure etc. There are severe side effects associated with atypical antipsychotics,

especially with widely used olanzapine, quetiapine and risperidone. Vitamin D and Vitamin E are

well known for their anti-oxidant activity. In our study we have emphasized the synergistic effects

of Vit D and Vit E administered with atypical anti psychotics in reducing the side effects and to

evaluate the improvement in the disease. For evaluation, Serum glutathione peroxidase (GPx) and

super oxide dismutase (SOD) were examined by colorimetric method. Tumor necrosis factor alpha

(TNF- $\alpha$ ) and interferon- $\gamma$  levels were analyzed by PCR whereas serum lipid profile was assessed

by commercially available kits. Improvement in illness was measured through Positive and

Negative Syndrome Scale score (PANSS)

We are in process of this clinical trial registration and would be happy to hear a positive

response.

Regards

Dr. M. Abid

Dr. Rabia Arshad